CLINICAL TRIAL: NCT05933564
Title: The Association Between Cognitive Reserve, Pain Catastrophizing, and Cognitive Function in Geriatric Patients With Chronic Pain: A Cross-sectional Study
Brief Title: Cognitive Reserve on Pain Catastrophizing and Cognitive Function in Geriatric Patients With Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/20265888
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Pain Patients with Varying Cognitive Reserve: Community-dwelling adults aged 65-85 years with chronic pain (≥3 months) attributable to osteoarthritis or neuropathic conditions.
  Interventions: Other: No intervention (cross-sectional study)

INTERVENTIONS:
Other: No intervention (cross-sectional study) — This is a cross-sectional study examining the association between cognitive reserve, pain catastrophizing, and cognitive function in geriatric patients with chronic pain; no intervention is being implemented or tested.

SUMMARY:
To investigate the association between cognitive reserve, pain catastrophizing, and cognitive function in geriatric patients with chronic pain, and to explore whether cognitive reserve moderates the relationship between pain catastrophizing and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 to 85 years
* Experiencing chronic pain (≥3 months) attributable to osteoarthritis or neuropathic conditions
* Able to read, write, and speak the language in which assessments are administered
* Willing and able to provide informed consent

Exclusion Criteria:

* Diagnosed with a neurodegenerative disorder (e.g., Alzheimer's disease, Parkinson's disease)
* History of significant head injury, stroke, or brain tumor
* Current substance abuse or dependence
* Severe psychiatric illness (e.g., schizophrenia, bipolar disorder)
* Significant sensory or motor impairments that may interfere with the ability to complete assessments

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of community-dwelling adults aged 65-85 years with chronic pain (≥3 months) attributable to osteoarthritis or neuropathic conditions.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Association between pain catastrophizing and cognitive function | Baseline assessment
  he relationship between pain catastrophizing, as measured by the Pain Catastrophizing Scale (PCS), and cognitive function, as measured by the Montreal Cognitive Assessment (MoCA version 7.1).

SECONDARY OUTCOMES:
Moderating effect of cognitive reserve on the association between pain catastrophizing and cognitive function | Baseline assessment
  Investigate whether cognitive reserve, as measured by the Cognitive Reserve Index Questionnaire (CRIq), moderates the relationship between pain catastrophizing (PCS) and cognitive function (MoCA version 7.1).

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No